CLINICAL TRIAL: NCT06251648
Title: Acute Lymphoblastic Leukaemia Related to Lenalidomide in Patients With Cancer: an Observational and Retrospective Study Using the WHO's Pharmacovigilance Database
Brief Title: Acute Lymphoblastic Leukaemia Related to Lenalidomide (LenALL)
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Pierre-Marie MORICE, PharmD, PhD, Dr, University Hospital, Caen
Other Study IDs: LenALL#01-02-2024
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lenalidomide — Patients exposed to LEN

SUMMARY:
Although lenalidomide (LEN) have proved effective in treating many cancers, few patients receiving LEN may experience rare but life-threatening adverse events such as Acute Lymphoblastic Leukaemia (ALL). Today, data about ALL are scarce.

The objective was to investigate reports of ALL adverse events related to LEN in patients with cancer using the World Health Organization (WHO) pharmacovigilance database.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO, also called VigiBase) at the time of the extraction
* Patients treated with at least LEN (L04AX04)

Exclusion Criteria:

-Chronology not compatible between LEN and ALL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated with LEN and experiencing ALL
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
ALL reports related to LEN (from WHO database). | From inception to February, 2024
  Identification of the ALL adverse events related to LEN reported in the World Health Organization (WHO) database of individual safety case reports.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No